CLINICAL TRIAL: NCT03142464
Title: Intravenous Fluids After Laparoscopic Cholecystectomy: Necessary or Dispensable. A Randomized Clinical Trial
Brief Title: Intravenous Fluids After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Professor of Surgery, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102908/2015
Record Dates: First submitted 2017-04-09; First posted 2017-05-05 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Nausea; Postoperative Vomiting; Renal Function Abnormal; Hunger; Thirst; Fluid Electrolyte Disorders
Keywords: saline solution; laparoscopy; cholecystectomy; outcomes
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Controls - convention postoperative IV fluids; intervention arm - no IV fluids postoperative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV fluids (No Intervention): Regular IV fluids (Glucose 5% and Sodium Chloride 10% or Ringer) at the surgeon description
- No IV fluids (Experimental): No IV fluids after the termination of the operation. T
  Interventions: Other: Suspension of the IV fluids

INTERVENTIONS:
Other: Suspension of the IV fluids — No IV fluids prescription, IV catheter filled with saline solution
  Arms: No IV fluids

SUMMARY:
Perioperative intravenous fluid (IV) administration has been the standard procedure since 1832 and, is a widely used practice sometimes under inadequate criteria. The present work aims at verifying the clinical need that justifies the common IV fluid prescription on the postoperative (PO) period in patients undergoing videolaparoscopic cholecystectomy (CVL) elective.

DETAILED DESCRIPTION:
Patients undergoing elective laparoscopy cholecystectomies were randomized to either routine practice fluid prescription (control group) or no IV fluids in the postoperative period. Thirst, hunger, presence of nausea and vomiting, renal function and personal satisfaction were assessed.

Body composition was evaluated by bioimpedance

ELIGIBILITY:
Inclusion Criteria: Elective laparoscopy cholescitectomy; no intraoperative complication -

Exclusion Criteria: Co-existing severe renal failure, cardiac failure or pulmonary disease

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Renal function | 24 hours
  Serum creatinine

SECONDARY OUTCOMES:
Presence of thirst | 24 hours
  Visual analog scale
Presence of nausea | 24 hours
  Visual analog scale
Total intravenous prescribed fluids per body weight | 24 hours

IPD SHARING:
Plan to Share IPD: No